CLINICAL TRIAL: NCT03513328
Title: PEDS024, Phase I/II Feasibility Study of Busulfan Fludarabine and Thiotepa Conditioning Regimen for Allogeneic Hematopoietic Stem-Cell Transplantation (HSCT) for Children With Non-Malignant Disorders
Brief Title: Conditioning Regimen for Allogeneic Hematopoietic Stem-Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Live Like Bella Pediatric Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201800798; PEDS024 (Other: UF Health); OCR17838 (Other: Universiy of Florida); AWD05935 (Other Grant/Funding Number: Live Like Bella Pediatric Cancer Research)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Bone Marrow Failure Syndrome; Thalassemia; Sickle Cell Disease; Diamond Blackfan Anemia; Acquired Neutropenia in Newborn; Acquired Anemia Hemolytic; Acquired Thrombocytopenia; Hemophagocytic Lymphohistiocytoses; Wiskott-Aldrich Syndrome; Chronic Granulomatous Disease; Common Variable Immunodeficiency; X-linked Lymphoproliferative Disease; Severe Combined Immunodeficiency; Hurler Syndrome; Mannosidosis; Adrenoleukodystrophy
Keywords: human leukocyte antigen (HLA)
MeSH Terms: conditions — Bone Marrow Failure Disorders; Thalassemia; Anemia, Sickle Cell; Anemia, Diamond-Blackfan; Anemia, Hemolytic; Lymphohistiocytosis, Hemophagocytic; Wiskott-Aldrich Syndrome; Granulomatous Disease, Chronic; Common Variable Immunodeficiency; Lymphoproliferative Disorders; Severe Combined Immunodeficiency; Mucopolysaccharidosis I; Mannosidase Deficiency Diseases; Adrenoleukodystrophy

STUDY DESIGN:
Intervention Model Description: The study builds in rules for escalation of thiotepa dose based on graft failure by day 42. Patients are stratified in two groups A (lower risk of graft failure) and B (higher risk of graft failure). Patients undergoing 10/10 HLA matched bone marrow and peripheral blood transplants are assigned to Group A, and patients receiving <10/10 matched bone marrow or peripheral blood, or receiving cord blood, even if fully matched, are assigned to Group B.
  If criteria for thiotepa dose escalation are met first in Group A, which has a lower risk of graft failure, thiotepa dose will be escalated for all subjects (Groups A and B). If criteria for thiotepa dose escalation are met first in Group B, dose will be escalated only in Group B and Group A will continue enrolling patients at a lower dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A--Thiotepa single dose (Experimental): Fully matched 10/10 subjects with lower risk of graft failure. Subjects will undergo 10/10 HLA (human leukocyte antigen) matched bone marrow and peripheral blood transplant. Subjects receive combination of single daily dose thiotepa (5 mg/kg) added to the backbone of targeted reduced dose IV busulfan, fludarabine and rabbit anti-thymocyte globulin (rATG).
  Interventions: Drug: Thiotepa--single daily dose
- Group A--Thiotepa escalated dose (Experimental): Fully matched 10/10 subjects with lower risk of graft failure. Subjects will undergo 10/10 HLA (human leukocyte antigen) matched bone marrow and peripheral blood transplant. Subjects receive combination of escalated dose of thiotepa (10 mg/kg) added to the backbone of targeted reduced dose IV busulfan, fludarabine and rabbit anti-thymocyte globulin (rATG).
  Interventions: Drug: Thiotepa--escalated dose
- Group B--Thiotepa single dose (Active Comparator): Subjects with higher risk of graft failure. Subjects will undergo transplant with <10/10 bone marrow or peripheral blood match, or receiving cord blood transplant. Subjects receive combination of single daily dose thiotepa (5 mg/kg) added to the backbone of targeted reduced dose IV busulfan, fludarabine and rabbit anti-thymocyte globulin (rATG).
  Interventions: Drug: Thiotepa--single daily dose
- Group B--Thiotepa escalated dose (Active Comparator): Subjects with higher risk of graft failure. Subjects will undergo transplant with <10/10 bone marrow or peripheral blood match, or receiving cord blood transplant. Subjects receive combination of escalated dose of thiotepa (10 mg/kg)added to the backbone of targeted reduced dose IV busulfan, fludarabine and rabbit anti-thymocyte globulin (rATG).
  Interventions: Drug: Thiotepa--escalated dose

INTERVENTIONS:
Drug: Thiotepa--single daily dose — Conditioning regimen for hematopoietic stem-cell transplant. Single daily IV dose of Thiotepa at 5 mg/kg.
  Arms: Group A--Thiotepa single dose; Group B--Thiotepa single dose
Drug: Thiotepa--escalated dose — Twice daily IV dose of Thiotepa at 5 mg/kg, twelve hours apart, 10mg/kg total.
  Arms: Group A--Thiotepa escalated dose; Group B--Thiotepa escalated dose

SUMMARY:
In this study, the investigators test 2 dose levels of thiotepa (5 mg/kg and 10 mg/kg) added to the backbone of targeted reduced dose IV busulfan, fludarabine and rabbit anti-thymocyte globulin (rATG) to determine the minimum effective dose required for reliable engraftment for subjects undergoing hematopoietic stem cell transplantation for non-malignant disease.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation is the only curative choice for a number of inherited bone marrow failure syndromes, hemoglobinopathies, metabolic disorders and primary immune deficiencies. While survival of these patients is typically better than survival of patients with malignancies, toxicities of conditioning regimens and failure of engraftment remain challenges. Most children with non-malignant disorders present with normocellular or even hypercellular bone marrow, posing a barrier to engraftment and requiring intensive conditioning. Commonly used backbone of busulfan and fludarabine, although well tolerated, results in variable engraftment, in particular with mismatched unrelated donors and cord blood recipients. In this study, the investigators test 2 dose levels of thiotepa (5 mg/kg and 10 mg/kg) added to the backbone of targeted reduced dose IV busulfan, fludarabine and rabbit anti-thymocyte globulin (rATG) in order to determine the minimum effective dose required for reliable engraftment. Subjects are stratified in groups A and B based the risk of graft failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses:

  * Hemoglobinopathies (e.g. thalassemia or sickle cell disease),
  * Cytopenias (e.g.Diamond-Blackfan anemia, congenital or acquired neutropenia, congenital or acquired thrombocytopenia, congenital or acquired anemia, and others, regardless clonality),
  * Hemophagocytic lymphohistiocytosis,
  * Primary immunodeficiencies (e.g. Wiscott Aldrich Syndrome, chronic granulomatous disease, common variable immune deficiency, X-linked lymphoproliferative disease, NK+ severe combined immune deficiencies),
  * Metabolic disorders (Hurler's syndrome, mannosidosis, adrenal leuko-dystrophy)
  * Other non-malignant disorders for which there is published evidence that HSCT (hematopoietic stem cell transplant) is a curative therapy.
* Donor Requirements

  * Related or unrelated donor who is suitable and willing to donate bone marrow or peripheral blood stem cells. HLA typing should be done by high-resolution typing at A, B, C, DrB1 and DQ loci and the donor should be at a minimum ≥8/10 match (with one antigen/allele mismatch allowed at A, B, or C-loci and other at DQ loci).
  * Cord blood units must be matched at a minimum of 6/8 antigens/alleles at A, B, C and DrB1 loci. High resolution typing at all loci is required. The minimum TNC dose pre-cryopreservation must be ≥3.7 x10^7/kg of recipient's weight, if a single cord blood unit is used, or at least 2x10^7/kg per unit, if two cord blood units are used. The mismatches cannot be at the same loci (e.g. double A mismatch).
  * Haploidentical related stem cell donor who is suitable and willing to donate peripheral blood stem cells. T-cell depletion is required if haploidentical donors are used. Pharmacologic GVHD prophylaxis will not be used for T-cell depleted transplant recipients.
* Adequate organ function defined as:

  * Cardiac: ejection fraction ≥55% or shortening fraction ≥30%
  * creatinine clearance ≥70 ml/min/1.73m2
  * Pulse oximetry >95% on room air or FEV1/DLCO >60%
  * LFTs < 3 x ULN, Total bilirubin <3 mg/dl (unless due to non-hepatic cause (e.g. Gilbert's syndrome or hemolysis)
* Lansky/Karnofsky score ≥60%
* Written informed consent obtained from the subject or parental/guardian permission ± child's assent per institutional guidelines
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy for at least 1 month after completion of conditioning. WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

  * Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
  * For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
  * Males with female partners of childbearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, or vasectomy) for at least one month after completion of conditioning.

Exclusion Criteria:

* Diagnoses that do not require myeloablative transplant for cure (e.g. NK- SCID patients), unless the subject previously did not engraft with non-myeloablative or reduced intensity conditioning transplant.
* Known or suspected sensitivity to chemotherapy or radiation (e.g Fanconi's anemia, Dyskeratosis congenita, Ligase IV deficiency, etc).
* Subjects with fast-progressing neurodegenerative disorders (e.g. Krabbe disease or adrenal leukodystrophy with Loes score of ≥10)
* Cytopenias with increased blasts (>5%)
* Presence of anti-donor HLA antibodies (positive anti-donor HLA antibody is defined as a positive cross-match test of any titer (by complement-dependent cytotoxicity or flow cytometric testing) or the presence of anti-donor HLA antibody to the high expression loci HLA-A, B, C, DRB1 with mean fluorescence intensity (MFI)>3000 by solid phase
* Prior allogeneic stem cell transplant, except for patients with immune deficiencies who underwent previous non-myeloablative or reduced intensity transplants.
* Haploidentical donor using in vivo T-cell depletion (e.g. post-transplant cyclophosphamide).
* Uncontrolled bacterial, viral, or fungal infection at the time of enrollment. Uncontrolled is defined as currently taking medication and with progression or no clinical improvement on adequate medical treatment.
* Seropositive for HIV
* Active Hepatitis B or C determined by a detectable viral load of HBV or HCV by PCR
* Bridging fibrosis or liver cirrhosis
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 1 months after the end of conditioning
* Females who are pregnant or breastfeeding
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Subjects demonstrating an inability to understand the study and comply with the study and/or follow-up procedures

Ages: 3 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2023-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Horn, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Children's Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from June 2018 through January 2021. Only Arm A enrolled patients due to change in clinical practice. No donors with HLA mismatch enrolled in this study.
Period: Overall Study
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Started | 6 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No enrollments in Group A Thiotepa escalated dose or Group B Arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose | Total
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 |  |  |  | 4
  Between 18 and 65 years | 2 |  |  |  | 2
  >=65 years | 0 |  |  |  | 0
Age, Continuous [Median (Full Range); unit: years] — Age at time of consent.
  years | 13 [0.5 to 24] |  |  |  | 13 [0.5 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 0 | 2
  Male | 4 | 0 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  | 0
  Not Hispanic or Latino | 6 |  |  |  | 6
  Unknown or Not Reported | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 2 |  |  |  | 2
  White | 4 |  |  |  | 4
  More than one race | 0 |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 |  |  |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Minimum Effective Dose (MED) of Thiotepa
Description: Assess the MED of thiotepa in combination with reduced-dose busulfan, fludarabine and rATG required to achieve engraftment in >90% subjects undergoing hematopoietic stem cell transplantation for non-malignant disorders.
Time Frame: Day 42
Population: MED dose of thiotepa in group A was determined to be 5 mg/kg in combination with Fludarabine and rATG. All six patients engrafted by day 42 using this dose. No subsequent escalation was done.
Measure: Number; unit: mg/kg
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
mg/kg | 5 |  |  |

2. Secondary Outcome: Percentage of Subjects With Graft Rejection/Failure.
Description: Percentage of all subjects who initiated conditioning regimen and have sustained engraftment failure.
Time Frame: Day 42; Day 365
Population: Risk of rejection was determined in Group A. None of the patients rejected the graft = 0% (95% CI 0-46%) either at Day 42 or Day 365
Measure: Number; unit: Percentage of participants
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Percentage of participants | 0 |  |  |

3. Secondary Outcome: Percentage of Subjects Without Disease Recurrence Who Are Alive at 24 Months Post Transplant
Description: Percentage of subjects who initiated conditioning regimen and are without evidence of underlying disease (DFS).
Time Frame: Month 24
Population: At 24 month OS and DFS was 100% (95% CI 54-100%) in group A, the OS and DFS could not have been evaluated for group B due to lack of enrollment
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Percentage of patients | 100 [54 to 100] |  |  |

4. Secondary Outcome: Percentage of Subjects Alive at 24 Months Post Transplant (OS)
Description: Percentage of subjects who initiated conditioning regimen and are alive at 24 months post transplant (OS).
Time Frame: Month 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Percentage of patients | 100 [54 to 100] |  |  |

5. Secondary Outcome: Evaluation of Transplant-related Mortality
Description: Percentage of subjects who initiated conditioning regimen and who died due to a cause unrelated to the underlying disease.
Time Frame: Month 12
Population: Transplant related mortality at 12 months post transplant was 0% (95% CI 0-46%) in Group A. Transplant-related mortality could not have been evaluated for group B due to lack of enrollment
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Percentage of patients | 0 [0 to 46] |  |  |

6. Secondary Outcome: Number of Participants With Grade 2-4 Acute Graft-versus-host Disease (GVDH)
Description: Graft-versus host disease symptoms measured using Modified Glucksberg Staging Criteria. (Scale 0-4; with 4 being most severe)
Time Frame: Month 12
Population: 1 of 6 patients developed GVHD grade 2-4.
Measure: Number; unit: Number of patients
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Number of patients | 1 |  |  |

7. Secondary Outcome: Percentage of Participants With Chronic Graft-versus-host Disease (cGVHD)
Description: Measures the frequency of chronic graft-vs-host disease in Group A participants
Time Frame: Month 24
Population: cGVHD in 2 of 6 participants
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Percentage of patients | 33 [0.4 to 78] |  |  |

8. Secondary Outcome: Percentage of Participants With Transplant-related Complications
Description: Complications gathered via CIBMTR (Center for International Blood & Marrow Transplant Research) post-transplant form was tabulated and described by treatment received.
Time Frame: 24 months
Population: Percentages of patient at risk for complications during first 2 years post transplant
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
Number analyzed (Participants) | 6 | 0 | 0 | 0
Percentage of patients
  Mucositis - 1st year post transplant | 100 [54 to 100] |  |  |
  Viral reactivations - first year post transplant | 67 [22 to 96] |  |  |
  Covid 19 Infection first year post transplant | 17 [0 to 64] |  |  |
  Bacterial Infection first year post transplant | 33 [0 to 78] |  |  |
  Hemorrhagic Cystitis in first year post transplant | 17 [0 to 64] |  |  |
  Viral reactivations in 2nd year post transplant | 67 [22 to 96] |  |  |
  Covid 19 infection in the 2nd year post transplant | 17 [0 to 64] |  |  |
  Bacterial Infections in the 2nd year post transplant | 17 [0 to 64] |  |  |

ADVERSE EVENTS:
Time Frame: First 100 days post transplant and AESI for 24 months.
Description: Grade III and higher adverse events and serious adverse events were monitored for first 100 days. All-Cause Mortality and AESI were monitored for 24 months.
Arm/Group | Group A--Thiotepa Single Dose | Group A--Thiotepa Escalated Dose | Group B--Thiotepa Single Dose | Group B--Thiotepa Escalated Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A--Thiotepa Single Dose (N=6) | Group A--Thiotepa Escalated Dose (N=0) | Group B--Thiotepa Single Dose (N=0) | Group B--Thiotepa Escalated Dose (N=0)
Mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Salmonella Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coag Negative Staph Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever and joint pain (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress secondary to mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tranaminitis (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to change in clinical practice, only patients with HLA matched donors were enrolled in this trial. Study was closed prematurely due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03513328/Prot_SAP_000.pdf